CLINICAL TRIAL: NCT06225180
Title: Review of Breast Abscess Management
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 021.TRA.2023.D
Record Dates: First submitted 2023-11-14; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Breast Abscess

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast abscesses are an unfortunate pathology that develop in patients, and treatment is often painful and unpleasant. The goal of this study is to identify risk factors associated with failure of aspiration as a primary intervention as opposed to incision and drainage in the hopes of adequately treating patients at initial presentation.

DETAILED DESCRIPTION:
The pendulum has now swung toward minimally invasive aspiration as the primary treatment modality, with multiple studies reporting superior cosmetic results. However, patients in these studies often required repeat breast aspirations, and sometimes ultimately required incision and drainage. Aspiration first for treatment of breast abscess may not be a wise choice for all patients if it results in increased antibiotic days, return to emergency department (ED)/increased cost, or prolonged pain from multiple procedures. Several studies have identified varying risk factors for aspiration failure as primary intervention for breast abscesses. More data is needed to confirm the true risk factors for failure.

ELIGIBILITY:
Inclusion Criteria:

* • ≥18 years of age

  * New diagnosis of N61.1 recorded in their Electronic Medical Record (EMR)

Exclusion Criteria:

* • <18 years of age

  * Pregnant
  * Incarcerated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years of age
  • New diagnosis of N61.1 recorded in their EMR
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2024-06-29 (Estimated); Study Completion 2024-06-29 (Estimated)

PRIMARY OUTCOMES:
Number of repeat interventions prior to resolution of abscess(s) | 5 years
  Determine the superiority of aspiration vs incision as primary intervention in treatment of breast abscesses

SECONDARY OUTCOMES:
Antibiotic days | 5 years
  number of days used antibiotics
Repeat aspiration | 5 years
  Frequency of aspiration
Return to Emergency Department ( ED) | 5 years
  Number of times of ED visit

CONTACTS AND LOCATIONS:
Overall Officials: Conner McDaniel, MD, Principal Investigator — Methodist Midlothian Medical Center
Locations (2):
- United States (2):
  - Clinical Research Institute at Methodist Health System, Dallas, Texas
  - Methodist Dallas Medical Center, Dallas, Texas